CLINICAL TRIAL: NCT05177640
Title: Early Prediction of Tumor Response to Treatment: Translation of 99mTc-Duramycin
Brief Title: Biodistribution and Dosimetry of 99mTc-Duramycin
Acronym: PicTURE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Molecular Targeting Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NIH 1R01CA226531 - 01A1
Record Dates: First submitted 2021-07-15; First posted 2022-01-04 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2021-07

CONDITIONS: Healthy Volunteers
Keywords: dosimetry, biodistribution, safety, 99mTc-duramycin
MeSH Terms: interventions — technetium 99m HYNIC-duramycin; Cell Death

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 99mTC-duramycin (Experimental): single dose of 99mTc-duramycin in healthy volunteers who will undergo SPECT-CT scanning at different time points
  Interventions: Drug: 99mTc-Duramycin

INTERVENTIONS:
Drug: 99mTc-Duramycin — This is a single dose study of 99mTc-duramycin in healthy volunteers who will undergo serial SPECT scanning
  Other Names: cell death

SUMMARY:
Conduct a first-in-human study in healthy volunteers to show safety, biodistribution and dosimetry of [99mTc]Duramycin.

DETAILED DESCRIPTION:
Monocenter, prospective microdosing study in healthy volunteers. Healthy volunteers will undergo a [99mTc]Duramycin whole-body planar and abdominal SPECT scan at different time points after one iv injection of the radiotracer (1 h, 2h, 3h, 6h and 24h), while vital signs, urine and faces analysis will be checked. Blood samples will be taken at 12 different time points: 9 blood samples for dosimetry study and 3 blood samples will be subjected to clinical laboratory chemistry (renal and liver function chemistry, hematology, and blood coagulation parameters).

ELIGIBILITY:
Inclusion Criteria:

* Males (n=4) or females (n=4) age 18 years or older
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Ability to give study-specific written informed consent.

Exclusion Criteria:

* Pregnant or lactating females (positive pregnancy test)
* Metal implants (e.g. pacemakers, osteosynthesis material)
* Body weight > 100 kg
* Severe claustrophobia
* Abnormal kidney or liver function tests
* Unable to comply with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Determine the biodistribution of [99mTc]Duramycin. | 24 hours
  Subjects will be dosed with 99mTc-Duramycin at Time 0 on Day 0, and a SPECT scan will be conducted immediately after the injection. Imaging will be repeated at 1 hour, 2 hours, 3 hours, 6 hours and 24 hours after dosing.
  All images generated will be reviewed for biodistribution.
Determine the dosimetry evaluation of [99mTc]Duramycin. | 24 hours
  Subjects will be dosed with 99mTc-Duramycin at Time 0 on Day 0, and a SPECT scan will be conducted immediately after the injection. Imaging will be repeated at 1 hour, 2 hours, 3 hours, 6 hours and 24 hours after dosing.
  All images generated will be reviewed for dosimetry.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0" | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sigrid Stroobants, prof, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Metelerkamp Cappenberg T, De Schepper S, Vangestel C, De Lombaerde S, Wyffels L, Van den Wyngaert T, Mattis J, Gray B, Pak K, Stroobants S, Elvas F. First-in-human study of a novel cell death tracer [99mTc]Tc-Duramycin: safety, biodistribution and radiation dosimetry in healthy volunteers. EJNMMI Radiopharm Chem. 2023 Aug 30;8(1):20. doi: 10.1186/s41181-023-00207-1. PMID 37646865